CLINICAL TRIAL: NCT04647396
Title: Biomarker- Guided Intervention to Prevent Acute Kidney Injury After Major Surgery. A Prospective Randomized Controlled Multicenter Trial (BigpAK-2)
Brief Title: Biomarker-guided Intervention to Prevent Acute Kidney Injury
Acronym: BigpAK-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 07-AnIt-20
Record Dates: First submitted 2020-10-12; First posted 2020-11-30 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Acute Kidney Injury
Keywords: biomarker
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Comprehensive Implementation of the Bundle recommended by the "Kidney Disease: Improving Global Outcomes Group" (KDIGO bundle)
- Control group (No Intervention)

INTERVENTIONS:
Other: Comprehensive Implementation of the Bundle recommended by the "Kidney Disease: Improving Global Outcomes Group" (KDIGO bundle) — Implementation of the KDIGO bundle for at least 12 hours
  1. discontinuation of all nephrotoxic drugs when possible
  2. optimization of volume status and hemodynamic parameters (consideration of a functional hemodynamic monitoring)
  3. close monitoring of serum creatinine, fluid balance and urinary output
  4. avoidance of hyperglycemia
  5. considerations of alternatives to radiocontrast agents
  6. discontinuation of angiotensin converting enzyme inhibitors and angiotensin receptor blockers in the perioperative period
  7. avoidance of HES, gelatin, and chlorid-rich solutions
  Arms: Intervention group

SUMMARY:
There is no specific therapy for acute kidney injury. It is presumed that supportive measures improve the care and outcome of patients with acute kidney injury. The investigators hypothesize that the implementation of a bundle of supportive measures adapted to patients undergoing major surgery reduces the occurrence of AKI.

This randomized prospective multicenter trial is needed to investigator whether the implementation of the bundle of measures is effective to prevent AKI in high risk patients undergoing major surgery.

DETAILED DESCRIPTION:
In earlier studies, interventions to treat acute kidney injury (AKI) were started after a functional damage of the kidneys was already established. However, none of the interventions had an effect in treating AKI. The Kidney Disease: Improving Global Outcomes (KDIGO) clinical practice guidelines recommend implementing different measures in patients at high risk for AKI, but the evidence that the implementation of the bundle (consisting of optimization of hemodynamics and perfusion pressure, avoidance of nephrotoxins and hyperglycemia) can prevent AKI is very weak. Biomarkers can be used to identify patients at high risk for AKI after surgery (prior to the development of AKI). The cell-cycle arrest biomarkers, Tissue Inhibitor of Metalloproteinases-2 (TIMP-2) and Insulin-like growth factor-binding protein 7 (IGFBP7), have been demonstrated to have the best predictive performance for the development of AKI after surgery as compared to other biomarkers. In addition, these biomarkers are not influenced by different co-morbidities or other clinical situations. In the BigpAK1 trial, which was a single-center trial, the authors investigated whether a biomarker-guided implementation of the KDIGO guidelines can reduce the occurrence of AKI in patients undergoing major non-cardiac surgery. The results demonstrate that the implementation of the KDIGO bundle in high risk patients for AKI ([TIMP-2]*[IGFBP7] between 0.3 and 2) significantly reduced the occurrence of AKI compared to the standard of care group. However, this was a single center trial which needs to be confirmed in a large trial. Therefore, based on these data, a definitive, prospective, randomized controlled, multicenter study including 1302 surgical patients at high risk for AKI identified by [TIMP-2]*[IGFBP7] will be performed.

The goal of this trial is to investigate the effect of the implementation of the KDIGO bundle in patients at high risk for AKI after major surgery compared to standard of care in the same patient population. This biomarker-guided approach (individualized therapy) enables to treat patients at high risk for AKI prior to a functional damage of the kidneys.

ELIGIBILITY:
Inclusion Criteria:

* Patients after major surgery who need to be admitted to the ICU
* Age > 18 years
* [TIMP-2]*[IGFBP7] ≥ 0.3 4-18 hours after surgery
* Inserted jugular central venous line and a urinary catheter
* Written informed consent.
* At least one additional risk factor for AKI

  1. Age > 75 years
  2. Critical illness such as ongoing requirement of vasopressor support and/or mechanical ventilation postoperatively
  3. Pre-existing chronic kidney disease (eGFR<60ml/min)
  4. Intraoperative use of radio contrast agents.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Pre- existing high stages of chronic kidney disease (stage 4 or 5 i.e. eGFR < 15 ml/ min)
* Kidney transplant within the last 12 month
* Known (Glomerulo-) Nephritis, interstitial nephritis or vasculitis
* Anuria at inclusion time
* Preexisting AKI
* Renal replacement therapy (RRT) within the last 90 days
* Indication for renal replacement at the time of inclusion
* Participation in another intervention trial that investigates a drug/intervention that affects kidney function
* Persons held in an institution by legal or official order
* Persons with any kind of dependency on the investigator or employed by the responsible institution or investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1180 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Occurence of moderate or severe AKI | 72 hours after start of intervention

SECONDARY OUTCOMES:
Adherence to the implementation of the KDIGO-bundle | 72 hours after start of intervention
  Number of patients in whom
  * Nephrotoxic agents were discontinued
  * Optimal volume status and perfusion pressure were ensured
  * The use of hemodynamic monitoring was considered
  * Serum creatinine and urine output were considered
  * Hyperglycemia was avoided
  * Alternatives to radiocontrast were considered
Severity of AKI | 3 days after start of intervention
  Severity of AKI as defined by the KDIGO guidelines based on creatinine or urine output parameter:
  Stage 1 Creatinine: 1.5-1.9 times baseline OR > 0.3 mg/dl (> 26.5 mmol/l) increase and/or urine output < 0.5 ml/kg/h for 6-12 hours
  Stage 2 Creatinine: 2.0-2.9 times baseline and/or urine output < 0.5 ml/kg/h for >= 12 hours
  Stage 3 Creatinine: 3.0 times baseline OR Increase in serum creatinine to >= 4.0 mg/dl (>= 353.6 mmol/l) OR Initiation of renal replacement therapy OR, In patients < 18 years, decrease in eGFR to < 35 ml/min per 1.73 m2 and/or urine output < 0.3 ml/kg/h for >= 24 hour
Changes in biomarker values | 12 hours after start of intervention
  Difference between the 12 h after initial measuring and the initial measuring [TIMP-2]*[IGFBP7] value
Free-days of mechanical ventilation | up to 3 days after start of intervention
Free-days of vasopressors | up to 3 days after start of intervention
Need of renal replacement therapy | up to 30 days after start of intervention
Need of renal replacement therapy | up to 90 days after start of intervention
Duration of renal replacement therapy | up to 30 days after start of intervention
Duration of renal replacement therapy | up to 90 days after start of intervention
Renal recovery | up to 90 days after start of intervention
  renal recovery is defined as complete recovery: serum creatinine levels < 0.5 mg/dl higher than baseline serum creatinine (creatinine level before surgery), partial recovery: serum creatinine > 0.5 mg/dl higher than baseline but not dialysis-dependence; non-recovery: patients who remained dialysis dependent
Mortality | 30 days after start of intervention
Mortality | 90 days after start of intervention
ICU and hospital stay | up to 90 days after start of intervention (until discharge)
Major adverse kidney events (MAKE) | up to 90 days after start of intervention
  - major adverse kidney events consisting of mortality, dialysis dependency persistent renal dysfunction (defined as serum creatinine ≥ 2x to baseline value at hospital discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Zarbock, MD, Study Chair — University Hospital Muenster, Dept. of Anesthesiology, Intensive Care Medicine and Pain Therapy
Locations (37):
- France (3):
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Service d´Anesthésie-Réanimation, Hôpital Edouard Herriot, Hospices Civils de Lyon, Lyon
  - Centre Hospitalier Universitaire de Reims, Reims
- Germany (13):
  - Department of Anaesthesiology and Intensive Care Medicine, Klinikum Bayreuth GmbH, Bayreuth
  - Department of Anesthesiology, Intensive Care Medicine and Pain Therapy, University Hospital Knappschaftskrankenhaus, Ruhr University Bochum, Bochum
  - Department of Anesthesiology and Intensive Care Medicine, University Hospital Bonn, Bonn
  - Department of Anesthesiology, Intensive Care and Pain Medicine, Klinikum Dortmund, Dortmund
  - Department of Anesthesiology and Intensive Care Medicine, University Hospital "Carl Gustav Carus", Technische Universität Dresden, Dresden
  - Department of Anesthesiology, University Hospital Düsseldorf, Heinrich-Heine-University Duesseldorf, Düsseldorf
  - Department of Anesthesiology and Intensive Care Medicine, University Hospital Essen, University Duisburg-Essen, Essen
  - Department of Anesthesiology, University Medical Center, Georg-August-University, Göttingen
  - Department of Anesthesiology, Heidelberg University Hospital, Heidelberg
  - Department of Anesthesiology and Intensive Care Medicine, Philipps-University, Marburg
  - Department of Anaesthesiology, Intensive Care and Pain Medicine, University Hospital, Münster
  - Department of Anesthesiology, Department of Anesthesiology and Critical Care, Franziskus Hospital Münster, Münster
  - Department of Anesthesiology and Intensive Care Medicine, University Hospital Tübingen, Eberhard Karls University Tübingen, Tübingen
- Italy (5):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - Department of Translational Medicine and for Romagna, St. Anne's Archbishop Hospital, University of Ferrara, Ferrara
  - Department of Health Sciences, Section of Anesthesiology, Intensive Care and Pain Medicine, University of Florence; Department of Anesthesia and Intensive Care, Section of Oncological Anesthesia and Intensive care, Azienda Ospedaliero Careggi, Florence
  - Santa Chiara Regional Hospital, APSS Trento, Trento
  - Department of Anesthesiology and Intensive Care, San Bortolo Hospital, Vicenza
- Department of Anaesthesiology, Laboratory of Experimental Intensive Care and Anaesthesiology (L.E.I.C.A.), Amsterdam UMC, Location Academic Medical Centre (AMC), Amsterdam, University of Amsterdam, Amsterdam, Netherlands
- Spain (9):
  - Department of Anaesthesiology and Intensive Care Medicine, Parc de Salut Mar, Barcelona
  - Hospital de Igualada, Barcelona
  - Department of Anesthesia and Perioperative Care, Infanta Leonor University Hospital, Madrid
  - Department of Anesthesiology, Hospital Universitario Ramón y Cajal, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Clínico San Carlos de Madrid, Madrid
  - Servicio de Anestesiologia y Reanimación, Hosp. Universitario de La Princesa, Madrid
  - Department of Anaesthesiology and Surgical Critical Care, Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen Macarena, Seville
- Adult Intensive Care Unit, Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland
- United Kingdom (5):
  - Centre for Experimental Medicine, School of Medicine, Dentistry, and Biomedical Sciences, Queen's University Belfast, Belfast
  - Intensive Care Unit, Royal Surrey County Hospital, Guildford
  - Department of Anaesthetics and Critical Care, Harefield Hospital, Harefield
  - Intensive Care Unit, Royal Liverpool University Hospital, Liverpool
  - Department of Critical Care, King's College London, Guy's & St Thomas' Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zarbock A, Ostermann M, Forni L, Bode C, Wild L, Putensen C, Roux DP, Martin EE, Arndt C, Rahmel T, de Rosa S, Monard C, Schneider AG, Glass A, Jung-Konig M, Romagnoli S, Gossage J, Lumlertgul N, Haaker JG, Ripolles-Melchor J, Spadaro S, Siniscalchi A, Futier E, Aupetitgendre L, Bhathal IR, Alvarez RG, Bernard A, Rosenberger P, Wempe C, Sadjadi M, Meersch M, Fischhuber K, Bellomo R, Kellum JA, von Groote T; BigpAK-2 study group. A preventive care strategy to reduce moderate or severe acute kidney injury after major surgery (BigpAK-2); a multinational, randomised clinical trial. Lancet. 2025 Dec 13;406(10521):2782-2791. doi: 10.1016/S0140-6736(25)01717-9. Epub 2025 Nov 13. PMID 41242333
- [Derived] von Groote T, Danzer MF, Meersch M, Zarbock A, Gerss J; BigpAK-2 study group. Statistical analysis plan for the biomarker-guided intervention to prevent acute kidney injury after major surgery (BigpAK-2) study: An international randomised controlled multicentre trial. Crit Care Resusc. 2024 Jun 21;26(2):80-86. doi: 10.1016/j.ccrj.2024.03.001. eCollection 2024 Jun. PMID 39072240
- [Derived] von Groote T, Meersch M, Romagnoli S, Ostermann M, Ripolles-Melchor J, Schneider AG, Vandenberghe W, Monard C, De Rosa S, Cattin L, Rahmel T, Adamzik M, Parise D, Candela-Toha A, Haaker JG, Gobel U, Bernard A, Lumlertgul N, Fernandez-Valdes-Bango P, Romero Bhathal I, Suarez-de-la-Rica A, Larmann J, Villa G, Spadaro S, Wulf H, Arndt C, Putensen C, Garcia-Alvarez R, Brandenburger T, Siniscalchi A, Ellerkmann R, Espeter F, Porschen C, Sadjadi M, Saadat-Gilani K, Weiss R, Gerss J, Kellum J, Zarbock A; BigpAK-2 Investigators. Biomarker-guided intervention to prevent acute kidney injury after major surgery (BigpAK-2 trial): study protocol for an international, prospective, randomised controlled multicentre trial. BMJ Open. 2023 Mar 27;13(3):e070240. doi: 10.1136/bmjopen-2022-070240. PMID 36972972

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT04647396/SAP_002.pdf